CLINICAL TRIAL: NCT05777486
Title: A Randomized Controlled Trial Examining How TikTok Influencers' Posts With Vs. Without Food Differentially Affect Youth Dietary Choices
Brief Title: Dietary and Cognitive Effects of Food Ads Posted by TikTok Influencers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 22-01632
Record Dates: First submitted 2023-03-08; First posted 2023-03-21 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Calorie Consumption
MeSH Terms: interventions — Food

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TikTok Influencer Ads with Food (Experimental): Participants randomized to view TikTok influencers' posts with food will view 4 ads associated with their condition and 2 filler ads, all of which are presented in counterbalanced order. They will report their reaction to the ads using the icons available on the TikTok platform (i.e. like, comment, or share). After viewing all of the TikTok ads, youth participants will complete the virtual snack selection task where they will see a virtual vending machine. All items will cost $2. Participants will be asked to select one snack and one beverage from the vending machine. After the snack selection task, participants will review the TikTok ads again and complete survey questions.
  Interventions: Behavioral: TikTok Ads - With Food
- TikTok Influencer Ads without Food (Experimental): Participants randomized to view TikTok influencers' posts without food will view 4 ads associated with their condition and 2 filler ads, all of which are presented in counterbalanced order. They will report their reaction to the ads using the icons available on the TikTok platform (i.e. like, comment, or share). After viewing all of the TikTok ads, youth participants will complete the virtual snack selection task where they will see a virtual vending machine. All items will cost $2. Participants will be asked to select one snack and one beverage from the vending machine. After the snack selection task, participants will review the TikTok ads again and complete survey questions.
  Interventions: Behavioral: TikTok Ads - Without Food

INTERVENTIONS:
Behavioral: TikTok Ads - With Food — TikTok posts from influencers promoting food.
  Arms: TikTok Influencer Ads with Food
Behavioral: TikTok Ads - Without Food — TikTok posts from influencers who are not promoting food.
  Arms: TikTok Influencer Ads without Food

SUMMARY:
Randomized and controlled experimental study to evaluate how influencer food ads on TikTok affect calorie purchases among youth (ages 10-13). Participants will be randomized to one of two conditions: (1) seeing an influencer with food or (2) seeing an influencer without food. Participants will complete a 15-minute survey in which they will be randomized to one of two conditions and view and rate TikTok influencer ads associated with their condition. Then they will complete a food purchasing task in which they will shop in an online store that will display six food items and six beverages. Finally, they will answer demographic questions (e.g., self-reported height and weight) and view a debriefing summary that describes the full purpose of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 10-13 years old
* Identify as only non-Latino White or only Black/African American
* Report that they log into TikTok at least once daily
* Read and speak English

Exclusion Criteria:

• Any criteria not met as listed above will bar an adolescent from participating in the study

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Calorie Count from Snacks Chosen at Virtual Vending Machine | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bragg, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Zora.hall@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Zora.hall@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.